CLINICAL TRIAL: NCT06593197
Title: Comparison Between Apremilast in Combination with NBUVB and NBUVB Alone in Vitiligo - a Randomized Controlled Trial
Brief Title: Efficacy and Safety of Apremilast in Combination with NBUVB and NBUVB Alone in Vitiligo Patients
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Madiha Sajid, Assistant Professor, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIMC/DUHS/DERMA/001/2024
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-01

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apremilast with phototherapy (Experimental)
- Phototherapy alone (Active Comparator)
  Interventions: Device: NB-UVB

INTERVENTIONS:
Combination Product: Apremilast with NB-UVB — Tab Apremilast 30 mg twice a day with NBUVB twice per week for 8 months
Device: NB-UVB — NBUVB only will be given twice per week for 8 months
  Arms: Phototherapy alone

SUMMARY:
Patients of non-segmental vitiligo, fulfilling the inclusion criteria will be selected from the OPD, dermatology department. It's an interventional study where Group A patient will be given NBUVB and Tab Apremilast 30 mg twice a day and Group B will receive NBUVB alone.

DETAILED DESCRIPTION:
Patients of non-segmental vitiligo, fulfilling the inclusion criteria will be selected from the OPD, dermatology department Dow university hospital. Informed consent will be obtained from all the patients.

Demographic details of patients including age, gender, education, occupation and marital status will be obtained. Further each patient will be asked about duration of vitiligo and any systemic medications used by the patients in the last 6 months will be recorded.

Body Surface Area will be calculated and patients with > 5% of BSA will be included in the study.

Subjects will be randomly divided by lottery method into two groups. Group A patients will be given NBUVB and Tab Apremilast 30 mg twice a day, and Group B patients will receive NBUVB alone.

Hematological baseline including CBC and LFTs will be advised to patients in Group A.

Vitiligo Area Severity Index (VASI) will be used to initially assess the patient at the baseline and later on to assess the regimentation in each of the patients of vitiligo on next 4 follow-ups. Each follow-up will be after every 8 weeks for a total of 32 weeks. CBC and LFTs will be repeated in Group A after 4 weeks of starting tab Apremilast 30 mg BD and then after 3 months. Any side effects seen during the study period will be recorded and managed accordingly DLQI Dermatological Life Quality Index (DLQI) questionnaire will be conducted with 30 vitiligo patients at the baseline and at the end of therapy.

All results will be collected and filled in proforma by the researcher. The results will be assessed statistically at the end of the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years and above
* Patients of both genders (male and female)
* Diagnosed patients of non-segmental vitiligo involving > 5% of BSA

Exclusion Criteria:

* Pregnant and lactating women
* Concomitant active infection like tuberculosis
* Personal history of cutaneous malignancy
* Use of apremilast in the past 4 weeks
* Use of phototherapy within 4 weeks before randomization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
To determine the frequency of patients halted their progression and extent of repigmentation | 32 weeks
  Halt in progression and extent of repigmentation from baseline to week 32 in both groups will be calculated by Scale named Vitiligo Area and Severity Index(VASI) done at the baseline and then at week 8, week 16, week 24 and 32.
  Score of the scale ranges from 0 -100 . Fall in the score will show the improvement.
To determine the frequency of patients showing decrease in the percentage of depigmented areas | 32 weeks
  This will be performed by calculating Body surface area (BSA ) at the baseline and at week 32 .
  The patient's palmar surface including their fingers = 1% BSA Scale grading is as follows, mild (less than 3%) moderate (3-10%) severe (greater than 10%)
  Fall in the percentage of depigmented area is taken as improvement .

SECONDARY OUTCOMES:
DLQI Score and Safety | 32 weeks
  Dermatology Life Quality Index (DLQI) score at week 32 compared to baseline Scale ranges from 0 to 30 0 - 1 no effect at all, 2 - 5 small effect, 6 -10 moderate effect , 11 - 20 very large effect, 21 - 30 extremely large effect on the life of patient.
  Decrease in the score will be a marker of improvement

OTHER OUTCOMES:
To determine the tolerability and safety of intervention | 32 weeks
  Documentation of Adverse Events during therapy

CONTACTS AND LOCATIONS:
Overall Officials: Principal DIMC, Study Chair — Dow International Medical college
Locations (1):
- Dow International Medical College , DUHS, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No